CLINICAL TRIAL: NCT06146296
Title: THE EFFECT OF VITAMIN C ON POST-ORTHODONTIC TREATMENT RELAPSE: A RANDOMIZED CONTROLLED CLINICAL TRIAL
Brief Title: THE EFFECT OF VITAMIN C ON POST-ORTHODONTIC TREATMENT RELAPSE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: #10/23
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Orthodontic Relapse

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intra-epidermal Vitamin C injection (Experimental)
  Interventions: Biological: Local Vitamin C injection
- Oral Vit-C supplement (Active Comparator)
  Interventions: Biological: Oral Vitamin C supplement
- Control group (No Intervention)

INTERVENTIONS:
Biological: Local Vitamin C injection — An injection of 1-1.5 ml of L-ascorbic acid, locally introduced in relation to the keratinized gingival tissues, with extension to the whole target region successively. The injected area will be massaged for equal distribution of the injected vitamin. Injections will be performed on the first day of retainer delivery (T0), after 1 month (T1), after 3 months (T2), and after 6 months (T3). Hence, a total of 4 local Vit-C injections will be performed over the study period.
  Arms: Intra-epidermal Vitamin C injection
Biological: Oral Vitamin C supplement — Patients will be prescribed a daily oral (systemic) Vit-C supplement to be taken over the follow up period.
  Arms: Oral Vit-C supplement

SUMMARY:
The aim of this study is to evaluate and compare the effect of locally injected and orally administered (systemic) Vitamin C on post-orthodontic treatment relapse

ELIGIBILITY:
Inclusion Criteria:

* Patients who were indicated for non-extraction orthodontic treatment.
* Adult patients with finished orthodontic treatment, using fixed appliance therapy.
* Patients with good oral hygiene, and a healthy periodontal condition.

Exclusion Criteria:

* Patients who received sectional fixed appliance therapy.
* Patients with hypodontia requiring tooth replacement in the retainer, as a temporary measure.
* Patients requiring fixed bonded retainers.
* Pregnant and lactating women.
* Patients with hereditary hemochromatosis.
* Cancer patients, receiving chemotherapy.
* Patients with chronic diseases such as diabetes, or those receiving drugs such as corticosteroids, both of which that may affect tooth movement.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of post-orthodontic relapse | up to 8 months
  Alginate impressions will be taken, and dental models will then be scanned using Sirona inEos X5 CAD/CAM lab scanner, producing 3D digital images of the dental models in the form of stereolithographic (STL) files, which will be subsequently imported into a computer software. Little's Irregularity Index (LII) will be employed for the measurement and the quantitative evaluation of the lower anterior segment alignment. The horizontal linear displacement of the anatomic contact points of each mandibular incisor from the adjacent anatomic point is measured, and the 5 displacements are then summed together. The summed value represents the degree of anterior irregularity as follows: 0 = Perfect alignment. 1-3 = Minimal irregularity. 4-6 = Moderate irregularity. 7-9 = Severe irregularity. 10 = Very severe irregularity.
Analysis of salivary alkaline phosphatase levels | up to 8 months
  Salivary samples will be collected and measured using chemical analysis. Rise in salivary alkaline phosphatase levels reflects inflammation and destruction of healthy tissues suggesting it as a clinical biomarker. The normal level of alkaline phosphatase is 20-140IU/L (international unit per liter) in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Samar M Adel, PhD, Principal Investigator — Alexandria University; Farah Y Eid, PhD, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt